CLINICAL TRIAL: NCT06321133
Title: High Flow Nasal Cannula Weaning in Acute Bronchiolitis - an Open-label Randomized Controlled Trials
Brief Title: High Flow Nasal Cannula Weaning in Acute Bronchiolitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Central Finland Hospital District (Other); Mikkeli Central Hospital (Other); Siun sote (Unknown)
Responsible Party: Principal Investigator, Ilari Kuitunen, Associate Professor, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5402589
Record Dates: First submitted 2024-02-13; First posted 2024-03-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Bronchiolitis
Keywords: Acute bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate ending (Experimental): High flow is ended immediately
  Interventions: Other: High flow nasal cannula immediate ending
- Weaning (Active Comparator): High flow is ended by gradually reducing the flow rate
  Interventions: Other: High flow nasal cannula weaning

INTERVENTIONS:
Other: High flow nasal cannula immediate ending — High flow is immediately ended
  Arms: Immediate ending
Other: High flow nasal cannula weaning — High flow is gradually weaned by reducing the flow rate
  Arms: Weaning

SUMMARY:
The goal of this clinical study is to compared two different strategies to end high flow nasal cannula treatment in acute bronchiolitis. This study compared the immediate ending of high flow treatment to weaning strategy, in which the flow rate is gradually decreased. The aim is to assess if the immediate ending shortens the hospitalization time and whether it is a safe strategy.

DETAILED DESCRIPTION:
Acute bronchiolitis is the most common cause of hospitalization among infants in Finland, with its primary etiology being the RS- virus. Acute bronchiolitis is defined in Finland as an infant's first respiratory distress before the age of 1. There is no effective pharmacological treatment for acute bronchiolitis. High-flow nasal cannula therapy has been shown in large randomized trials to reduce the risk of intensive care unit admission for children. High-flow nasal cannulas are typically used at a flow rate of 2 liters per kilogram per minute. Despite widespread use, there is insufficient evidence to determine whether high-flow therapy should be discontinued abruptly or gradually tapered. Observational studies indicate that the majority of units opt for abrupt discontinuation. Common criteria for discontinuation include weaning off supplemental oxygen and maintaining normal oxygenation on room air for 4-6 hours. Gradual weaning has been shown in observational studies to prolong hospitalization compared to immediate cessation of therapy. In a randomized controlled trial conducted in a pediatric intensive care unit, direct discontinuation shortened the duration of treatment by up to two days. However, there have been no previous randomized trials conducted on bronchiolitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed acute bronchiolitis
* High flow nasal cannula treatment has lasted for at least 12 hours
* Measured saturation 95 or more with room air
* High flow rate is maximum 2l/kg/min
* The treating doctors considers the infant suitable to be without high flow

Exclusion Criteria:

* Major congenital anomaly of lungs, hearts or diaphragm
* Bacterial pneumonia
* Parents do not give consent

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalization time from randomization | One week
  Time in hours from the randomization to the time the family leaves hospital.

SECONDARY OUTCOMES:
Treatment failures | One week
  Need to restart the high flow therapy
Readmission rate | Seven days from discharge
  Need for readmission
Overall hospitalization time | One week
  The overall time, which includes the time interval prior to randomization

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Siun Sote, Joensuu
  - Central Finland Hospital District, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Mikkeli Central Hospital, Mikkeli

IPD SHARING:
Plan to Share IPD: No